CLINICAL TRIAL: NCT01270412
Title: Platelet Rich Plasma (PRP) as a Treatment for Knee Osteoarthritis - A Randomized-Double-Blind Trial
Brief Title: Platelet Rich Plasma (PRP) as a Treatment for Knee Osteoarthritis PRP as a Treatment for Knee Osteoarthritis
Acronym: PRP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Dr. Lior Laver, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMC10196-2010CTIL
Record Dates: First submitted 2010-12-20; First posted 2011-01-05 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; PRP; PRGF; Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Intercellular Signaling Peptides and Proteins; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platelet Rich Plasma (Preparation Rich in Growth Factors) (Experimental): intra articular injection 6ml of platelet-derived preparation rich in growth factors
  Interventions: Biological: Platelet Rich Plasma (Preparation Rich in Growth Factors)
- Hyaluronic acid (Active Comparator): Drug: hyaluronic acid 20 mg / 2 ml Other Name: Arthrease
  Interventions: Biological: Platelet Rich Plasma (Preparation Rich in Growth Factors); Drug: Hyaluronic acid

INTERVENTIONS:
Biological: Platelet Rich Plasma (Preparation Rich in Growth Factors) — intra articular injection 6ml
  Other Names: Platelet-derived preparation rich in growth factors
Drug: Hyaluronic acid — Intra articular injections: 20 mg / 2 ml
  Other Names: "Arthrease"
  Arms: Hyaluronic acid

SUMMARY:
Autologous platelet-secreted growth factors (GFs) may have therapeutic effects in osteoarthritis (OA) capsular joints via multiple mechanisms. The aim is to examine the effect of a platelet-derived preparation rich in growth factors (PRGFs) in OA of the knee.

DETAILED DESCRIPTION:
Autologous platelet-secreted growth factors (GFs) may have therapeutic effects in osteoarthritis (OA) capsular joints via multiple mechanisms. The investigators aim is to examine the effect of a platelet-derived preparation rich in growth factors(PRGFs) in OA of the knee, using parameters of pain, function, quality of life and safety.

ELIGIBILITY:
Inclusion Criteria:

* age 40-75 years old
* diagnosed Oa of the knee more then 1 year
* no knee deformation

Exclusion Criteria:

* mental of physical disabilities
* pregnancy
* deformities of the knee

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in pain, function, quality of life and activity level in knee osteoarthritis | 1 -2 years
  Improvement in pain, function, quality of life, activity level - using scores adapted to measure these parameters in knee osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Laver, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel